CLINICAL TRIAL: NCT03267108
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Escalation and Verification Clinical Study to Assess the Safety and Efficacy of Pulsed Inhaled Nitric Oxide (iNO) in Subjects at Risk of Pulmonary Hypertension Associated With Pulmonary Fibrosis on Long Term Oxygen Therapy (Part 1 and Part 2) - REBUILD
Brief Title: A Study to Assess Pulsed Inhaled Nitric Oxide in Subjects With Pulmonary Fibrosis at Risk for Pulmonary Hypertension
Acronym: REBUILD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial did not meet its primary endpoint, hence was terminated due to futility.
Sponsor: Bellerophon Pulse Technologies (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-PHPF-001
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: Pulmonary Fibrosis; PF; Pulmonary Hypertension; Inhaled Nitric Oxide; iNO; Long Term Oxygen Therapy; Oxygen; REBUILD; INOpulse; pulsed inhaled nitric oxide; fILD; fibrotic interstitial lung disease; portable pulsed inhaled nitric oxide
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Inhaled Nitric Oxide (iNO) (Active Comparator): Pulsed inhaled iNO 45 mcg/kg Ideal Body Weight (IBW)/hour (hr)
  Interventions: Combination Product: INOpulse®
- Placebo (Placebo Comparator): Pulsed inhaled N2, 99.999% gas
  Interventions: Combination Product: Placebo
- Open Label Extension (Other): Pulsed inhaled iNO 45 mcg/kg IBW/hr
  Interventions: Combination Product: Open Label Extension

INTERVENTIONS:
Combination Product: INOpulse® — Subjects will be treated by means of an INOpulse® device using an INOpulse® nasal cannula.
  Arms: Inhaled Nitric Oxide (iNO)
Combination Product: Placebo — Subjects will be treated by means of an INOpulse® device using an INOpulse® nasal cannula.
  Arms: Placebo
Combination Product: Open Label Extension — Subjects will be treated by means of an INOpulse® device using an INOpulse® nasal cannula.
  Arms: Open Label Extension

SUMMARY:
A randomized, double-blind, placebo-controlled dose escalation and verification study to assess the safety and efficacy of pulsed inhaled nitric oxide (iNO) in subjects at risk for pulmonary hypertension associated with pulmonary fibrosis on long term oxygen therapy (Part 1 and Part 2) - REBUILD

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled dose escalation and verification clinical study to assess the safety and efficacy of pulsed inhaled nitric oxide (iNO) in subjects at risk for pulmonary hypertension associated with pulmonary fibrosis on long term oxygen therapy (Part 1 and Part 2) - REBUILD

ELIGIBILITY:
Inclusion criteria:

* A high resolution CT scan performed in the 6 months prior to screening associated with one of the following conditions and confirmed using guidelines, as per American Thoracic Society (ATS) / European Respiratory Society (ERS) / Japanese Respiratory Society (JRS) / Latin American Thoracic Association (ALAT):

  * Major IIPs (idiopathic interstitial pneumonias) diagnosis or suspected as one of the following:

    * Idiopathic pulmonary fibrosis
    * Idiopathic nonspecific interstitial pneumonia
    * Respiratory bronchiolitis-interstitial lung disease
    * Desquamative interstitial pneumonia
    * Cryptogenic organizing pneumonia
    * Acute interstitial pneumonia
  * Rare IIPs diagnosis by one of the following:

    * Idiopathic lymphoid interstitial pneumonia
    * Idiopathic pleuroparenchymal fibroelastosis
  * Unclassifiable idiopathic interstitial pneumonias

    * Chronic hypersensitivity pneumonitis
    * Occupational lung disease
  * Connective Tissue Disease associated with IPF (CTD-ILD)
  * Interstitial Pneumonia with Autoimmune Features (IPAF)
* Have been using oxygen therapy by nasal cannula for at least 4 weeks (including use limited to exertion)
* 6MWD ≥ 100 meters and ≤ 400 meters at screening and Baseline/Randomization visits.
* World Health Organization (WHO) Functional Class II-IV
* Forced Vital Capacity ≥ 40% predicted within the 60 day Screening period
* Age between 18 and 80 years (inclusive) at screening

Exclusion criteria:

* For women of child-bearing potential: Pregnant or breastfeeding females at Screening, or planning to get pregnant, or unwilling to use appropriate contraception if sexually active to avoid pregnancy during the study and for at least 30 days after discontinuation of the study drug.
* Heart failure with reduced ejection fraction (HFrEF; systolic heart failure) with an ejection fraction of < 40%; or severe HF with preserved EF (HFpEF; diastolic HF)
* History of sarcoidosis
* History of chronic thrombo-embolic pulmonary hypertension (CTEPH; WHO group 4 PH)
* Smoking within 3 months of Screening and/or unwilling to avoid smoking throughout the study
* Body mass index (BMI) >40 kg/m2 at screening
* Intermittent uncontrolled atrial fibrillation, in the opinion of the Principal Investigator
* Known severe hepatic impairment, in the opinion of the Principal Investigator
* Known severe renal impairment (Chronic Kidney Disease Epidemiology Collaboration (CKDEPI) 2009 equation [Levy 2009] calculated creatinine clearance <30 ml/min) at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) as Measured by Actigraphy | Baseline to Month 4
  Part 1 - Blinded Treatment Period
Adverse Events and Serious Adverse Events with Long Term INOpulse Therapy | Baseline to Month 4
  Part 2 - Open Label Extension (OLE)

SECONDARY OUTCOMES:
Change in Overall Activity as Measured by Actigraphy | Baseline to M4
  Part 1 - Blinded Treatment Period
Change in University of California San Diego (UCSD) Shortness of Breath Questionnaire (SOBQ) | Baseline to Month 4
  Part 1 Blinded Treatment Period: The UCSD SOBQ is a 24-item questionnaire developed to measure breathlessness associated with activities of daily living, on a scale between zero and five where 0 is not at all breathless and 5 is maximally breathless or too breathless to do the activity. The responses to all items are summed up to provide the overall score that can range from 0 (best outcome) to 120 (worst outcome).
Change in St. George Respiratory Questionnaire (SGRQ) - Activity, Impacts & Total | Baseline to Month 4
  Part 1 Blinded Treatment Period: SGRQ is a tool for assessing quality of life that has previously been validated for the use with patients with interstitial lung disease. It is a responsive tool that has three domains: symptoms, activity and impact (on daily life)
Time to Clinical Worsening | Baseline to Month 4
  Part 1 - Blinded Treatment Period
Time to Clinical Deterioration | Baseline to Month 4
  Part 1 Blinded Treatment Period
Time to Clinical Improvement | Baseline to Month 4
  Part 1 Blinded Treatment Period
Change in 6 Minute Walk Distance | Baseline to Month 4
  Part 1 Blinded Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, Study Director — Bellerophon Therapeutics
Locations (64):
- United States (61):
  - University of Alabama, Birmingham, Alabama
  - Banner - University Medical Center Arizona, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of California San Francisco, Fresno, California
  - University of California, Los Angeles, California
  - Amicis Research, Northridge, California
  - Paloma Medical Group, Paloma, California
  - University of California Davis Health, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - UC Denver Anschutz Medical Center, Aurora, Colorado
  - National Jewish, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - St. Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - University of Miami, Miami, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Piedmont Healthcare, Austell, Georgia
  - Northwestern, Chicago, Illinois
  - North Shore University Hospital, Evanston, Illinois
  - Loyola University, Maywood, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Ascension St. Vincent Hospital, Indianapolis, Indiana
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - Atlantic Health Respiratory Institute, Summit, New Jersey
  - NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - The University of North Carolina at Chapel Hill Marsico Clinical Research Center, Chapel Hill, North Carolina
  - Pulmonix, LLC/LeBauer Cone Health, Greensboro, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Thomas Jefferson University Korman Respiratory Institute, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Metroplex Pulmonary and Sleep, McKinney, Texas
  - University of Utah Health Sciences, Salt Lake City, Utah
  - Inova Heart and Vascular Institute Advanced Lung Disease Clinic, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Queen's University/Hotel Dieu Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nathan SD, Rajicic N, Dudenhofer R, Hussain R, Argula R, Bandyopadhyay D, Luckhardt T, Muehlemann N, Flaherty KR, Glassberg MK, Lancaster L, Raghu G, Fernandes P. Inhaled Nitric Oxide in Fibrotic Lung Disease: A Randomized, Double-Blind, Placebo-controlled Trial. Ann Am Thorac Soc. 2024 Dec;21(12):1661-1669. doi: 10.1513/AnnalsATS.202406-662OC. PMID 39141673